CLINICAL TRIAL: NCT03497468
Title: Effects of Task-oriented Training on Functional Mobility and Fatigue in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Kamer Unal, Lecturer, PhD, PT, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: kunal
Record Dates: First submitted 2018-04-03; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: task-oriented training; exercise training; mobility; balance; fatigue; quality of life
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients in this group will receive combined exercise training included aerobic and strengthening exercises, 3 times a week for 6 weeks. All exercise sessions will be performed under the supervision of a physiotherapist.
  Interventions: Other: Combined exercise training
- Training group (Experimental): Patients in this group will receive task-oriented training additional to combined exercise training 3 times a week for 6 weeks. Task-oriented training included more functional daily life mobility activities like reaching, obstacle walking, stairs climbing. All exercise sessions will be performed under the supervision of a physiotherapist.
  Interventions: Other: Task-oriented training

INTERVENTIONS:
Other: Combined exercise training — Aerobic training with cycle ergometer %60-80 of maximal Heart Rate, submaximal level, strengthening of the major muscles of upper and lower extremities
  Arms: Control group
Other: Task-oriented training — Functional reaching, walking on different obstacles and floor,sitting and standing on different levels and surface,walking around obstacle, climbing stairs with different height and surface
  Arms: Training group

SUMMARY:
Multiple Sclerosis (MS) is inflammatory, demyelinating and autoimmune disease of the central nervous system. It is usually seen with relapses and genetic and environmental factors play a role in the etiology. Neurological symptoms seen in MS restrict the patient's daily activity and social role participation. Mobility problems and fatigue are the most important reasons of role limitations and decreased quality of life. The importance of exercise training in disease management has been emphasized in recent years. However, few studies have investigated the effects of task-oriented trainings on symptoms of the disease. The aim of this sudy is to investigate the effects of task-oriented training additional to combined exercise training on functional capacity, mobility, balance, fatigue and quality of life in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis diagnosis
* Expanded Disability Status Scale > 5,5
* No cognitive problems
* No relapses in the last 3 months
* No other neurological or chronic disease

Exclusion Criteria:

* Relapse during the intervention
* Exercise intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | 6 weeks
  Change from baseline functional capacity with six minute walking test

SECONDARY OUTCOMES:
dynamic gait skills | 6 weeks
  Change from baseline functional mobility with dynamic gait index
limitation of gait | 6 weeks
  Change from baseline functional mobility with MS walking scale-12
dynamic balance and fall risk | 6 weeks
  Change from baseline functional mobility with timed up and go test
sitatic balance | 6 weeks
  Change from baseline balance with functional reach test
dynamic balance | 6 weeks
  Change from baseline balance with berg balance scale
severity of fatigue | 6 weeks
  Change from baseline fatigue with fatigue severity scale
impact of fatigue | 6 weeks
  Change from baseline fatigue with fatigue impact scale
Quality of life | 6 weeks
  Change from baseline quality of life with MS quality of life instrument-54

IPD SHARING:
Plan to Share IPD: Undecided